CLINICAL TRIAL: NCT05833074
Title: Evaluating the Efficacy of Annual CHTC Retesting Among Male Couples at High Risk of HIV Infection
Acronym: 4Us Part B
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Tyrel Starks, Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01 DA050508-S1; R01DA050508-03S1 (NIH)
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Counseling; chitinase C

STUDY DESIGN:
Intervention Model Description: Participants are randomized (with equal allocation) to either couples HIV testing and counseling retesting or an individual HIV testing control.
Who Masked: Outcomes Assessor
Masking Description: Research assistants are not given access to information about study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couples HIV testing and counseling retesting (Experimental): Couples HIV testing and counseling is completed following Centers for Disease Control and Prevention (CDC) standard protocol. Participants also complete any adjunct CHTC components associated with their originally assigned condition in NCT05000866.
  Interventions: Behavioral: Couples HIV testing and counseling
- Individual HIV testing (Active Comparator): Individual HIV testing and counseling.
  Interventions: Behavioral: Individual HIV testing and counseling

INTERVENTIONS:
Behavioral: Couples HIV testing and counseling — Couples HIV testing follows a CDC published protocol for delivery of HIV testing to relationship partners. HIV test results are obtained from Oraquick (FDA approved for at home HIV testing)
  Other Names: CHTC
  Arms: Couples HIV testing and counseling retesting
Behavioral: Individual HIV testing and counseling — Individual HIV testing and counseling uses a counseling protocol based on the standard of care for routine HIV pre- and post-test counseling. HIV test results are obtained from Oraquick (FDA approved for at home testing)
  Other Names: HTC
  Arms: Individual HIV testing

SUMMARY:
This randomized controlled trial evaluates the efficacy of couples HIV testing and counseling retesting. Eligible couples previously enrolled in NCT05000866 are invited to participate. Those who do are randomized to either couples HIV testing and counseling (CHTC) retesting or an individual HIV testing control. Follow-ups occur 3 and 6 months post intervention.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the benefits associated with couples HIV testing and counseling (CHTC) resting. After their 12-month follow-up, those participants who remain in the same relationship they were in at the time of their baseline will be offered the opportunity to continue in the components proposed in this revision. Those who consent will be randomized to either complete a second session of CHTC or to a comparison condition in which both partners receive a routine individual HIV test. HIV positive partners in serodiscordant couples randomized to the control condition will receive information about anti-retroviral treatment adherence and U=U (undetectable = untransmissible). Given potential attrition and rates of relationship dissolution, we anticipate randomizing 200 couples (80% of the original sample). Follow-up assessments will be conducted 3 and 6 months after retesting (15 and 18 months after the participants' original baseline appointment).

ELIGIBILITY:
Inclusion:

1. enrolled previously in the parent study DA050508 (NCT05000866).
2. in a relationship with the same main partner with whom they completed the baseline intervention session.
3. both partners in the couple must consent to continue with activities specified in this revision.
4. completion of the 12-month assessment associated with participation in the parent study prior to consenting to participate in activities specified under this revision.

Exclusion: any of the following at the 12-month follow-up:

1. serious psychiatric symptoms;
2. current suicidal/homicidal ideation;
3. gross cognitive impairment
4. a history of severe physical or sexual Intimate Partner Violence (IPV) victimization in the current relationship.

Ages: 17 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — cismale
Enrollment: 384 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
number of condomless anal sex acts with a casual partner in the absence of PrEP | 6 months
  Number of total anal sex acts (insertive and receptive) with casual partners reported on quarterly timeline follow-back assessments

SECONDARY OUTCOMES:
Binge drinking | 6 months
  Number of days on which 5 or more drinks containing alcohol were reported on the quarterly timeline follow-back interview
pre-exposure prophylaxis (PrEP) uptake | 6 months
  self-reported receipt of a PrEP-prescription
PrEP adherence | 6 months
  taking 4 or more doses weekly as prescribed reported on quarterly timeline follow-back assessments
Drug use Frequency | 6 months
  Number of reported days of illicit drug use (amphetamines, cocaine/crack, gama hydroxybutyric acid (GHB), ketamine or ecstasy) reported on quarterly timeline follow-back assessments

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Hunter College, New York, New York

IPD SHARING:
Plan to Share IPD: No
Participant-level data will be shared upon request and at the discretion of the study PI under the terms of a memorandum of understanding signed by officials at the transmitting and receiving institutions.

REFERENCES:
- [Derived] Starks TJ, Kyre K, Castiblanco J, Parker JN, Kahle E, Stephenson R, Cain D. Comparing Repeated (Annual) Couples HIV Testing and Counseling to Individual HIV Testing and Counseling Among Male Couples at High Risk of HIV Infection: Protocol for a Randomized Control Trial. JMIR Res Protoc. 2024 Feb 13;13:e53023. doi: 10.2196/53023. PMID 38349737